CLINICAL TRIAL: NCT04095442
Title: Effect of Antibacterial Mouthwash on Muscle Function in Healthy Young Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Coggan, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1907204336
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Quadriceps Muscle
Keywords: muscle power; nitric oxide; muscle speed; oral microbiome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cepacol (Active Comparator)
  Interventions: Device: Cepacol
- Tom's Natural Mouthwash (Sham Comparator)
  Interventions: Device: Tom's Natural Mouthwash

INTERVENTIONS:
Device: Cepacol — Twice-daily use of Cepacol per the manufacturer's guidelines
  Arms: Cepacol
Device: Tom's Natural Mouthwash — Twice-daily use of Tom's Natural Mouthwash per the manufacturer's guidelines
  Arms: Tom's Natural Mouthwash

SUMMARY:
The purpose of this study is to determine the effects of antibacterial mouthwash on muscle speed and power in healthy young men and women. We have previously demonstrated that drinking beetroot juice, a source of dietary nitrate and therefore nitric oxide, increases muscle function in this population. Antibacterial mouthwash has been shown to interfere with the conversion of dietary nitrate to nitric oxide. We therefore hypothesize that it will diminish nitric oxide bioavailability and inhibit muscle contractility.

DETAILED DESCRIPTION:
Study Visit One:

During an initial visit, subjects will complete the informed consent process, be instructed on the requirements of the study, and practice the exercise protocol (see below).

Study Visit Two:

Subjects will be tested after they have avoided exercise, caffeine, alcohol, chewing gum, and foods high in nitrate (e.g., spinach, beets, collard greens) for at least 24 hours. They will also be asked to not use any mouthwash products during this period. They will then provide provide a saliva sample for subsequent measurement of nitrate and nitrite concentrations and have their breath nitric oxide levels measured using a portable analyzer. The maximal knee extensor speed and power of their knee extensor muscles will then be measured using an isokinetic dynamometer. This machine can control the speed of movement while measuring the maximal force (torque) that a subject can voluntarily produce.

Subjects will then be randomly assigned to receive either an antibacterial mouthwash (Cepacol©, Reckitt Benckiser, Parsippany, NJ) or, as a control solution, an alcohol-free "natural" mouthwash (Tom's of Maine©, Kennebunk, ME). Participants will be asked to rinse their mouth as directed on the product's packaging for 30 s twice per day for 7 (+/-2) days and to record the usage of the mouthwash on a provided form. Subjects will then return for Study Visit 3 (see below). This is considered a single-blind study, which means that the investigators will not know what type of mouthwash a subject is receives.

Study Visit Three:

At the end of the treatment period, subjects will be asked to return to undergo the same procedures as described for Study Visit Two.

ELIGIBILITY:
Inclusion:

* Men and Women age 18-30 years old
* No current use of mouthwash

Exclusion:

* Men and Women <18 or 30> y of age
* Unable to provide informed consent
* Current users of mouthwash
* Current antibiotic use
* Current smokers
* Currently pregnant or lactating
* Stage II hypertension (resting blood pressure >140/>90)

An answer of yes to any of the seven questions on the first page of the Physical Activity Readiness Questionnaire (PAR-Q) indicating that the subject is not physically ready for exercise without a medical exam. These exclusions include the following:

* If participant's doctor has ever said that he/she has a heart condition and that he/she should only do physical activity recommended by a doctor
* Pain in chest when doing physical activity
* In past month, chest pain when not doing physical activity
* If participant has ever lost balance because of dizziness or has ever lost consciousness
* Bone or joint problem that could be made worse by change in physical activity
* Currently on prescribed drugs for blood pressure or heart condition.
* If the participant knows of any other reason why he/she should not do physical activity.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Health and Human Sciences, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cepacol | Tom's Natural Mouthwash
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cepacol | Tom's Natural Mouthwash | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (4) | 23 (3) | 22 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Muscle Function
Description: Maximal knee extensor speed determined using isokinetic dynamometry
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 13 | 13
rad/s | 11.0 (2.2) | 13.1 (2.5)

2. Primary Outcome: Muscle Function
Description: Maximal knee extensor speed determined using isokinetic dynamometry
Time Frame: 7 day
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 13 | 13
rad/s | 13.3 (3.0) | 13.6 (2.8)

3. Secondary Outcome: Salivary Nitrate
Description: Salivary concentration of nitrate
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 13 | 13
umol/L | 407 (229) | 595 (359)

4. Secondary Outcome: Salivary Nitrite
Description: Salivary concentration of nitrite
Time Frame: 7 day
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 13 | 13
umol/L | 602 (490) | 533 (310)

5. Secondary Outcome: Breath Nitric Oxide
Description: Breath nitric oxide level
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 8 | 7
ppm | 17 (10) | 20 (9)

6. Secondary Outcome: Breath Nitric Oxide
Description: Breath nitric oxide level
Time Frame: 7 day
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Cepacol | Tom's Natural Mouthwash
Number analyzed (Participants) | 8 | 7
ppm | 17 (7) | 20 (10)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Cepacol | Tom's Natural Mouthwash
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04095442/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04095442/ICF_001.pdf